CLINICAL TRIAL: NCT02566174
Title: Family Caregiving Role Adjustment and Dyadic Mutuality: A Mixed Methods Study
Brief Title: Family Caregiving Role Adjustment and Dyadic Mutuality
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999915206; 15-CC-N206
Record Dates: First submitted 2015-10-01; First posted 2015-10-02 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-09-18

CONDITIONS: Family Caregiver and Patient Mutual Negotiation of Roles and Responsibilities
Keywords: Cancer Caregivers; Cancer Patients; Role Adjustment; Mutuality; Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

Cancer causes changes in the lives of patients and in the lives of their caregivers. Patients and caregivers feel stress and they affect each other as they deal with these changes. They each cope with cancer diagnosis and treatment on their own. They also cope together. Researchers want to explore this shared change of roles and responsibilities. They will do this by gaining insight into the social experience of cancer caregiving. They also want to better understand the ways caregiver/patient teams manage the cancer diagnosis and experience. This can help find new ways to support caregivers and their patients.

Objective:

To explore the shared change of roles and responsibilities of patients and caregivers by studying the social experience of cancer caregiving.

Eligibility:

English speakers ages 18 and older who are one of the following:

A cancer patients at the NIH Clinical Center (CC)

A caregiver of a CC cancer patient

Design:

Participants will have been screened by the CC.

Patients and caregivers will be interviewed separately. This will last up to an hour and a half.

Participants will complete online surveys.

Participants may have a follow-up phone interview. This will last up to 15 minutes.

DETAILED DESCRIPTION:
Family caregiving is recognized as a significant public health problem, with approximately 66 million adult family caregivers in the United States providing services valued at an estimated $450 billion per year. These individuals are considered informal caregivers, in contrast to formal, paid caregivers such as nurses. Family caregivers suffer role strain and burden of caring that increases their risk for morbidity and mortality, which is the reason why they have been the focus of much caregiver research in recent decades. Improving health outcomes for family caregivers of cancer patients has involved developing approaches to reduce stress by boosting caregiver preparedness, mastery, and self-efficacy; however, in recent years there has been a progressive shift in the way the cancer caregiving experience has been characterized. This characterization has moved away from a focus on the individual to a focus on the caregiver-patient dyad. This shift has occurred, in part, because research has shown that each person in the dyad impacts the way in which the other person adjusts to his/her new role and responsibilities. Thus, the way this occurs is important since these adjustments not only influence the health of the dyadic relationship but also impact the couple s overall well-being.

Current focus on mutual or dyadic coping with cancer diagnosis and treatment stems from the understanding that caregivers and patients work individually, but also together to manage their shared stress and to make meaning out of their mutual experience. Because of this, mutuality and interdependence in dyadic coping extend beyond social support. Dyads collaborate, negotiate, and problem-solve to jointly manage stress and make decisions related to a diagnosis such as cancer. However, there has been little systematic inquiry into the dynamics of shared role adjustment in the cancer family caregiving dyad even though the stress of chronic illness appears to affect both the patient and the caregiver s well-being. The social experience of managing an illness such as cancer and the adjustments made to accommodate the new life situation are the first steps in what is often a prolonged disease trajectory that will require many other changes and transitions along the way.

Therefore, the primary objective for this study conducted in phase one is to explore family caregiver and care recipient mutual negotiation of roles and responsibilities by gaining insight into the social experience of cancer family caregiving that will have application to practice and guide further study. Phase two is contingent upon sample size, with the goal to further explore quantitative measures of individual caregiver and patient as well as dyadic well-being with regard to role adjustment and mutuality. A particular focus will be on dyads who are flourishing and those who are collaborating, to determine what they are doing differently.

A convergent parallel mixed methods study will be conducted using a grounded theory approach to data collection and analysis. A purposive sample of cancer patient participants and their designated family caregiver will be recruited from the National Institutes of Health Clinical Center. Final sample size will depend on conceptual and theoretical saturation, with an anticipated sample to include approximately 20 caregiver-patient dyads. A focused interview guide with open ended questions and probes will be used. During data collection and analysis, data will be compared to previous interviews and to the literature so that gaps in the developing framework can be identified and questions for subsequent interviews adjusted. To capture the experiences and perceptions of the interviewee, interviews with caregivers and care recipient participants will be conducted separately and by the same researcher. During analysis, both interviews will be analyzed on the level of the patient, of the family caregiver, and of the dyadic interaction (e.g. of categories and themes) between the two. Participants will also complete a socio-demographic questionnaire, Neuro QoL Ability to Participate in Social Roles and Activities, and Satisfaction with Social Roles and Activities-Short Forms, the Family Caregiving Inventory for Mutuality Scale, and the Mental Health Continuum-Short Form. This quantitative data will be triangulated and merged with conceptual categories from the caregiver and the care recipient interviews and will be used to compare subgroups to further illuminate qualitative findings.

Sacrifices caregivers make can lead to burden and stress, or to positive adjustment and growth. Through a better understanding of role adjustment and dyadic mutuality, we believe it will be possible to identify novel ways to support caregivers and their patients as they cope day to day and look toward the future.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patient participants will be recruited if they are at least 18 years of age, have a cancer diagnosis and are a patient at the NIH Clinical Center. They must be at least 6 weeks from the end of active treatment, be in a cancer caregiving situation with a spouse, partner (including non-traditional partner), significant other, family member or friend, be able to read and write English, and participate in a verbal interview (either face to face or by phone).

Caregiver Participants will be identified by the patient as the most involved in caregiving and therefore most likely the designated caregiver. The dyadic relationship will be co-defined and co-confirmed by both parties based on the researcher s understanding of dyadic dynamics. Caregiver participants will also be at least 18 years of age, be a spouse or partner (including non-traditional partner), significant other, family member or friend, be involved in the cancer caregiving situation with the care recipient for at least 6 months, be able to read and write English, and be able to participate in a verbal interview (either face to face or by phone).

EXCLUSION CRITERIA:

Patient participants will be excluded if under age 18, are not fully aware of diagnosis and treatment, if they are not a spouse or partner , (including non-traditional partner), significant other, family member or friend, if they are unable to participate in a verbal interview (either face to face or by phone) or are unable to read

or write English. A patient who has enrolled with one caregiver cannot enroll with another caregiver. A single caregiver must be identified for the duration of the protocol.

Caregiver Participants will be excluded if they are under age 18, are not the designated person identified by the care recipient as being most involved in their care, and if they are not a spouse or partner , (including non-traditional partner), significant other, family member or friend, if they are unable to participate in a verbal interview (either by face to face or by phone), or are unable to read or write English.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10-01; Primary Completion 2017-08-24 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Role Adjustment | on-going for Phase I
  by gaining insights into the social experience of cancer family caregiving that will have application to practice and guide further study
Mutuality | on-going for Phase I
  by gaining insights into the social experience of cancer family caregiving that will have application to practice and guide further study

SECONDARY OUTCOMES:
Patient and caregiver mutuality effect on patient well-being | 9/1/2017
Patient and caregiver mutuality effect on caregiver well-being | 9/1/2017

CONTACTS AND LOCATIONS:
Overall Officials: Margaret F Bevans, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Badr H, Carmack CL, Kashy DA, Cristofanilli M, Revenson TA. Dyadic coping in metastatic breast cancer. Health Psychol. 2010 Mar;29(2):169-80. doi: 10.1037/a0018165. PMID 20230090
- [Background] Park EO, Schumacher KL. The state of the science of family caregiver-care receiver mutuality: a systematic review. Nurs Inq. 2014 Jun;21(2):140-52. doi: 10.1111/nin.12032. Epub 2013 Apr 26. PMID 23617406
- [Background] Gibbons SW, Ross A, Bevans M. Liminality as a conceptual frame for understanding the family caregiving rite of passage: an integrative review. Res Nurs Health. 2014 Oct;37(5):423-36. doi: 10.1002/nur.21622. Epub 2014 Aug 30. PMID 25176315